CLINICAL TRIAL: NCT06225076
Title: A Randomized Controlled Study to Explore the Effect of Stellate Ganglion Block in Dysphagic Patients With Bulbar Palsy After Ischemic Stroke
Brief Title: Efficacy of Stellate Ganglion Block in Dysphagic Patients With Bulbar Palsy After Ischemic Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0112
Record Dates: First submitted 2024-01-13; First posted 2024-01-25 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Bulbar Palsy
MeSH Terms: conditions — Bulbar Palsy, Progressive | interventions — Lidocaine; Injections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The observation group (Experimental): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 20 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Procedure: Stellate ganglion block; Drug: Lidocaine Hydrochloride
- The control group (Active Comparator): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 20 days.
  Interventions: Behavioral: Comprehensive rehabilitation

INTERVENTIONS:
Behavioral: Comprehensive rehabilitation — All the participants are provided with the comprehensive rehabilitation (routine rehabilitation and swallowing function training). The routine rehabilitation included intervention for risk factors (blood pressure, blood lipids, blood glucose, smoking and alcohol restriction, exercise, etc.).
  Regrading swallowing function training, both groups are given swallowing function training, including 1) exercises of closure of the vocal folds, pharyngeal, and laryngeal muscles exercises, and respiratory muscle strength training, for 15 min each time and twice per day. 2) isotonic／isometric swallowing exercises, supraglottic swallowing exercises, for 20 min each time and twice per day. 3) effortful swallowing exercises, and cough reflex training, for 10 min each time and twice per day.
Procedure: Stellate ganglion block — the patients in the observation group were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: The observation group
Drug: Lidocaine Hydrochloride — the patients in the observation group were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Other Names: Injection
  Arms: The observation group

SUMMARY:
This is a randomized controlled study, including dysphagic patients with bulbar palsy after ischemic stroke who were received in the department of rehabilitation medicine in 3 hospitals in China. All patients are randomly allocated to the observation group or the control group. Both groups are provided with comprehensive rehabilitation. Besides, the observation group additionally undergoes the stellate ganglion block. At admission and after 20-day treatment, video fluoroscopic swallowing study, and penetration-aspiration scale, Functional Oral Intake Scale, Flexible laryngoscope are used to assess swallowing function.

DETAILED DESCRIPTION:
Palliation of dysphagia in patients with bulbar palsy after ischemic stroke continues to be a challenge.This is a randomized controlled study, including dysphagic patients with bulbar palsy after ischemic stroke who were received in the department of rehabilitation medicine in 3 hospitals in China. All patients are randomly allocated to the observation group or the control group. Both groups are provided with comprehensive rehabilitation. Besides, the observation group additionally undergoes the stellate ganglion block. At admission and after 20-day treatment, video fluoroscopic swallowing study, and penetration-aspiration scale, Functional Oral Intake Scale, Flexible laryngoscope are used to assess swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic stroke according to the diagnostic criteria, with the stroke occurring in the medulla oblongata and diagnosed as bulbar palsy.
* Upper Esophageal Sphincter did not open or opened ineffectively, with food residue or aspiration, revealed by Videofluoroscopic Swallow Study.
* Age >18 years.
* First-time stroke.
* Steady vital signs,
* Transferred or admitted to the Department of Rehabilitation Medicine within 15d after onset.

Exclusion Criteria:

* The bulbar palsy caused by other diseases, such as neurodegenerative diseases.
* Pseudobulbar palsy.
* Complicated with other neurological diseases.
* Tracheostomy tube inserted.
* Simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.
* Dysphagia caused by other possible diseases.
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 20
  On the day 1 and day 20, Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. As the level increased, the severity of dysphagia also increased.

SECONDARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 20
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.
Video Fluoroscopic Swallowing Study | day 1 and day 20
  Video Fluoroscopic Swallowing Study, which is considered as the "gold standard", swallowing process is divided into four periods: cognitive, oral, pharyngeal, and esophageal periods with a total score of 10 and a higher score indicates better swallowing ability (less dysphagia).
Murray secretion severity scale | day 1 and day 20
  Murray secretion severity scale is used for assessment of Pharyngeal secretion. The result was divided into 0-3 levels (0, normal; 1, a small amount of secretion remained and not entering the laryngeal vestibule; 2: temporary accumulation in the laryngeal vestibule; 3: persistent accumulation in the laryngeal vestibule. A higher score indicates the worse dysphagia.
Yale pharyngeal residue severity rating scale | day 1 and day 20
  The Yale pharyngeal residue severity rating scale was recruited for assessment of Pharyngeal residue.The result would be divided into 5 levels (1, no residue; 2, the covered pharyngeal mucosa; 3, mild residue, less than 50%; 4, moderate residue, more than 50%; 5, severe residue, spillage from laryngeal vestibule observed). A higher score indicates the worse dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng Da First Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No